CLINICAL TRIAL: NCT02180139
Title: Optimizing tDCS in Cervical Dystonia
Brief Title: tDCS in Cervical Dystonia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was withdrawn due to lack of funding and staff availability.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDCS-2014
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Primary motor cortex (M1) stimulation (Experimental): Treatment by transcranial direct current stimulation will be targeted to the motor cortex for all treatment sessions with Bilateral M1 with cathode to contralateral M1 and anode to ipsilateral M1, 15 minutes (Goal: decrease contralateral M1 excitability)
  Interventions: Device: transcranial direct current stimulation
- Cerebellum stimulation (Experimental): Treatment with transcranial direct current stimulation will be targeted to the cerebellum at every session with anode to ipsilateral cerebellum with cathode to ipsilateral side of face, 15 minutes (Goal: increase ipsilateral cerebellum activation which exerts inhibitory effect on motor circuits)
  Interventions: Device: transcranial direct current stimulation
- Combined M1 and Cerebellum stimulation (Experimental): Treatment with transcranial direct current stimulation will be placed with M1 anode contralateral + cerebellum anode. M1 will first be 'primed' with anode on contralateral M1, cathode on face, for 10 min, followed immediately by 15 min of cerebellar stimulation as in #2. (Goal: prime the contralateral M1 with increased excitability to engage a potentially larger effect from the following ipsilateral cerebellar stimulation that will be excited to exert inhibitory effect on the motor circuits including M1)
  Interventions: Device: transcranial direct current stimulation
- Sham stimulation (Placebo Comparator): transcranial direct current stimulation will be given in placebo form. Sham stimulation: electrode placement will be same as M1. Sham tDCS will be applied by ramping down current intensity to 0 after 30 seconds following standard practice for sham tDCS.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — tDCS using a constant current of 2 mA via two 35 cm2 saline soaked sponge electrodes. Treatment is 1x/day for 4 days.
  Other Names: Transcranial Technologies; TCT Research Limited, Kowloon, Hong Kong

SUMMARY:
Dystonia is a devastating disorder defined by involuntary, sustained muscle contractions or abnormal postures that can affect any part of the body. Cervical dystonia (CD) is the most pervasive form of dystonia affecting 60-90,000 individuals in the United States alone and is characterized by involuntary twisting of the neck. The symptoms of CD are disabling, disfiguring, painful, and have a strongly negative impact on quality of life, including social withdrawal and depression. At present, there is no treatment that has been shown to have long term benefit in CD. Standard of care (SOC) is botulinum toxin, which temporarily paralyzes affected muscles, resulting in reduced muscle spasms. This treatment has many undesirable side effects, variable effectiveness, is expensive, and must be repeated every 3 months throughout the lifespan. Physical therapy based treatments aimed at retraining posture or stretching dystonic muscles are largely ineffective and not typically delivered as a part of standard of care. There is an urgent need for novel and effective therapies. Emerging technologies, specifically non-invasive brain stimulation (NBS), have demonstrated compelling evidence to make a meaningful impact in the lives of people with CD. In this study, individuals with cervical dystonia will be randomly assigned to receive tDCS for 15 minutes daily for 4 days in 1 of 4 stimulation location groups.

Hypothesis 1: One location of stimulation will result in clear benefit with at least 1 standard deviation (SD) improvement in the CDQ-24, the primary outcome measure, at 1-week follow-up.

Hypothesis 2: The cortical silent period will be the most sensitive measure investigated and will demonstrate significant increase in inhibition as determined by an elongation of silent period in the affected upper trapezius muscle.

Hypothesis 3: The stimulation location determined to be most effective in Objective 1 will produce the greatest physiologic change in inhibition increase.

Hypothesis 4: The hypothesis for this aim is if certain characteristics can predict response to treatment, a strong association will be seen between baseline measure(s) and the primary outcome measure. A thorough assessment of characteristics including: age, sex, duration of symptoms, genotyping for two specific polymorphisms, botulinum toxin history, baseline measures of outcome variables, measures of brain excitability, and genetic testing will predict response.

DETAILED DESCRIPTION:
Study Purpose

This study will investigate the use of an experimental research device called transcranial direct current stimulation (tDCS). tDCS is a way to stimulate the brain with potential therapeutic benefits. It works by either increasing or decreasing brain excitability. This is done by delivering a current to the outside of the head. This weak electrical current then passes through the skull and modulates the underlying brain tissue. Genetic factors may contribute to the effectiveness of this intervention; therefore, a saliva sample will be collected to assess the status of two genes: Brain derived neurotrophic factor (BDNF) and apolipoprotein E4. Our purpose is to determine the best location of stimulation for tDCS that improves the symptoms and quality of life in people with CD. The results of this study will help to identify alternative interventions for people with cervical dystonia. Brain excitability will be measured using an additional form of non-invasive brain stimulation, specifically by a device called a transcranial magnetic stimulator. By applying a magnetic field to the outside of the head, electrical currents are produced within the brain that can transiently affect brain activity and be recorded though electrodes on your skin. Using this procedure, different areas of the brain can be studied to gain a greater understanding of the brain physiology in patients with cervical dystonia.

Procedures

Intervention: Briefly, non-invasive brain stimulation can be delivered safely and painlessly via different mechanisms with the goal of either exciting or inhibiting the underlying brain issue. In focal dystonia, as indicated above, there is thought to be a lack of inhibition, thus settings are typically used to increase inhibition. Transcranial direct current stimulation (tDCS) is one device that has been shown to be safe and effective at modulating excitation and inhibition in humans and has been used extensively in a variety of research applications for over 10 years. In addition to the potential physiologic benefit of altering excitability, tDCS is a particularly practical technique for use in people with CD, because it does not require one's head to remain still, thus not applying additional stress to the impaired neck.

An investigator will deliver tDCS using a constant current of 2 milliamps (mA) using a direct current stimulator (TCT Research Limited, Hong Kong) via two 35 cm2 saline soaked sponge electrodes. Treatment is 1x/day for 4 days. Electrode placement will be at one of four locations referenced in terms of dystonic head-turn resting position (i.e. if head turns to the left, the primary muscles involved are on the left, so contralateral M1 would be the right hemisphere): 1) Bilateral M1 with cathode to contralateral M1 and anode to ipsilateral M1, 15 minutes (Goal: decrease contralateral M1 excitability); 2) Cerebellum with anode to ipsilateral cerebellum with cathode to ipsilateral side of face, 15 minutes (Goal: increase ipsilateral cerebellum activation which exerts inhibitory effect on motor circuits); 3) M1+cerebellum: M1 will first be 'primed' with anode on contralateral M1, cathode on face, for 10 min, followed immediately by 15 min of cerebellar stimulation as in #2. (Goal: prime the contralateral M1 with increased excitability to engage a potentially larger effect from the following ipsilateral cerebellar stimulation that will be excited to exert inhibitory effect on the motor circuits including M1); or 4) Sham stimulation: electrode placement will be same as M1. Sham tDCS will be applied by ramping down current intensity to 0 after 30 seconds following standard practice for sham tDCS (Gandiga et al. 2006).

Pre-testing (Day1) will occur 10 weeks post standard care (SC) visit, so the participant will be near most impaired level of functioning prior to 12 week visit for botulinum (BTX) injection. tDCS will be delivered on day 1 and each subsequent day for 4 days. Posttesting will occur on Day5 and then 1 week later prior to SC visit (follow up- day 12). The primary endpoint of interest is follow up at one week.

Cortical Excitability Testing: Before and after intervention, single-pulse TMS will be delivered with a figure of eight coil (90 mm wing diameter) (MagStim Co., Whitland, Dyfed, Wales), positioned over M1. The 'hotspot' over the M1 contralateral to the direction of dystonic head turn will be used to collect motor evoked potentials (MEPs) in cervical muscles (upper trapezius) ipsilateral to head turn will be located and marked on the scalp. Various measures will be collected according to established methods to assess cortical excitability by single and paired pulse TMS.

Clinical assessment: Severity of CD will be assessed before and after the intervention. Behavioral measures will be administered by an investigator, blinded to intervention and will be assessed pre and post each intervention and at follow up. The primary endpoint of interest is the Craniocervical Dystonia Questionnaire CDQ-24. This primary outcome was selected because it is a patient-rated, disease-specific assessment of quality of life, which we feel should be the primary issue of concern. Secondary measures are TWSTRS and visual analog scale.

CDQ-24: The CDQ-24 contains 24 items with 5 subscales: stigma, emotional well-being, pain, activities of daily living and social/family life. Internal consistency and reliability is satisfactory for all sub-scales and total score with good sensitivity and high test/retest reliability (Muller, 2004).

TWSTRS. Toronto Western Spasmodic Torticollis Rating Scale is an outcome measure used to rate severity, disability and pain in CD (Consky et al., 1990). TWSTRS utilizes three sub-scores of physician-based severity (0-35), patient-based disability (0-30) and pain (0-20) with higher scores indicating greater severity of symptoms. Inter-observer reliability is excellent (rs=99) and good for disability and pain measurements (r˃0.88). The global severity scale was moderate (rs=0.63)(Salvia et al., 2006). TWSTRS exam will be videotaped for posthoc assessment by investigator blinded to group and testing period.

Visual Analog Scale (VAS). At the end of each intervention session participants will be asked to rate the ease of movement and perceived pain during cervical rotation in the contralateral direction to their head turn using VAS for self-assessment.

Adverse reactions. Adverse reactions will be recorded using established reporting forms.

Genetic Testing: At the last session, a saliva sample will be collected for genetic screening for BDNF and apolipoprotein E4 polymorphisms. We will collect approximately 2 ml (less than one-half teaspoon) of saliva by asking the subject to spit into a tube. It may take up to 30 minutes to provide a saliva sample, however, most people typically require less time (approximately 5 minutes). Collection of saliva using Oragene Discover is non-invasive and there are no anticipated personal risks of injury.

ELIGIBILITY:
Inclusion Criteria:

1. 21-65 years of age
2. Segmental dystonia, defined as dystonia in the neck plus another region is allowed, but CD must be primary source of disability.
3. Medications for dystonia are allowed, but they must be on a stable dose for the duration of the experiment. Individuals may be receiving BTX injections, but must be on a 2-cycle stable dose prior to experiment (first SC visit). Individuals who do not take BTX are also allowed to participate.

Exclusion Criteria:

1. Any surgical intervention or musculoskeletal impairment that would interfere with participation (eg., neck fusion, deep brain stimulation, peripheral denervation)
2. secondary dystonia (eg., Parkinson syndrome)
3. any neurologic or psychiatric disability that would interfere with participation
4. pregnancy
5. history of seizure within the last two years

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Cervical Dystonia Questionnaire (CDQ-24) | up to Day 6
  This primary outcome was selected because it is a patient-rated, disease-specific assessment of quality of life, which we feel should be the primary issue of concern.

SECONDARY OUTCOMES:
Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) | Day 1, Day 5, Day 6
  Toronto Western Spasmodic Torticollis Rating Scale is an outcome measure used to rate severity, disability and pain in CD. TWSTRS utilizes three sub-scores of physician-based severity (0-35), patient-based disability (0-30) and pain (0-20) with higher scores indicating greater severity of symptoms. Inter-observer reliability is excellent (rs=99) and good for disability and pain measurements (r˃0.88). The global severity scale was moderate (rs=0.63). TWSTRS exam will be videotaped for posthoc assessment by investigator blinded to group and testing period.
Visual Analog Scale (VAS) | Day 1, Day 5, Day 6
  At the end of each intervention session participants will be asked to rate the ease of movement and perceived pain during cervical rotation in the contralateral direction to their head turn using VAS for self-assessment.
Cortical Excitability as measured by transcranial magnetic stimulation | Day 1, Day 5, Day 6
  Single and paired pulse testing to assess GABAergic and glutaminergic network function

OTHER OUTCOMES:
Adverse reactions | Day 1, Day 2, Day 3, Day 4 (all days with intervention)
  Adverse reactions will be recorded using established reporting forms.
Genetic Testing | Day 6
  At the last session, a saliva sample will be collected for genetic screening for BDNF and apolipoprotein E4 polymorphisms. We will collect approximately 2 ml (less than one-half teaspoon) of saliva by asking the subject to spit into a tube. It may take up to 30 minutes to provide a saliva sample, however, most people typically require less time (approximately 5 minutes). Collection of saliva using Oragene Discover is non-invasive and there are no anticipated personal risks of injury.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa J Kimberley, PT, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Background] Muller J, Wissel J, Kemmler G, Voller B, Bodner T, Schneider A, Wenning GK, Poewe W. Craniocervical dystonia questionnaire (CDQ-24): development and validation of a disease-specific quality of life instrument. J Neurol Neurosurg Psychiatry. 2004 May;75(5):749-53. doi: 10.1136/jnnp.2003.013441. PMID 15090572
- [Background] Consky, E. S., Basinski, A., Belle, L., Ranawaya, R., & Lang, A. E. (1990). The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS): assessment of validity and inter-rater reliability. Neurology, 40(suppl 1), 445.
- [Background] Salvia P, Champagne O, Feipel V, Rooze M, de Beyl DZ. Clinical and goniometric evaluation of patients with spasmodic torticollis. Clin Biomech (Bristol). 2006 May;21(4):323-9. doi: 10.1016/j.clinbiomech.2005.11.011. Epub 2006 Jan 19. PMID 16427167